CLINICAL TRIAL: NCT03844659
Title: A Randomized Controlled Trial of Playing "The Most Relaxing Song in the World" During Labor Epidural Placement and Its Effects on Anxiety and Satisfaction
Brief Title: Music's Effects on Anxiety During Epidural Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, David Gutman, Principal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00078958
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Anxiety; Satisfaction
MeSH Terms: conditions — Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The song "Weightless" by Marconi Union will be playing during subjects labor epidural placement.
  Interventions: Other: Song "Weightless" by Marconi Union
- Non Intervention Group (Other): No song will be played during subjects labor epidural placement.
  Interventions: Other: No Song

INTERVENTIONS:
Other: Song "Weightless" by Marconi Union — Patients will be randomized to the intervention group (the song "Weightless" by Marconi Union will be playing) during subjects labor epidural placement. The intervention in this study is solely the addition of music.
  Arms: Intervention Group
Other: No Song — No song will be played during subjects labor epidural placement.
  Arms: Non Intervention Group

SUMMARY:
The objective of the study is to determine if playing the song "Weightless" by Marconi Union during labor epidural placement, decreases laboring parturient anxiety and improves satisfaction with the experience.

ELIGIBILITY:
Inclusion Criteria

* Females ages 18 years and older committed to delivery by the obstetrical team (natural labor or induction of labor)
* English speaking
* Able to give informed consent
* Having an epidural placed Exclusion Criteria
* Patient refusal
* Intrauterine fetal demise
* Imminent delivery
* Existing music use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant females
Enrollment: 100 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Mean Score of Anxiety Before Epidural Placement | Immediately prior to procedure
  3 different measures of anxiety prior to the procedure based on the State Trait Anxiety Inventory: 1) Numeric Rating Scale from 0-10 with 0 representing no anxiety and 10 representing worst anxiety possible. 2) Asking patient response to the question "Are you calm" with options scaling from "very much, moderately, somewhat, or not at all". 3) Asking the patient to answer the question "are you relaxed?" with options scaling from "very much, moderately, somewhat, or not at all." "Very much" will be treated as a positive finding and "moderately, somewhat, or not at all" as negative. The short form of the State Trait Anxiety Inventory with these three measures has been shown to be a reliable measure of anxiety. A fourth measure used will be a Visual Analog Scale from 0-100 of overall anxiety with 0 representing no anxiety and 100 representing the worst anxiety possible.
Mean Score of Anxiety After Epidural Placement | Immediately after procedure
  As soon as the epidural has been placed and appropriate documentation for the procedure is completed, both groups will take the same surveys again.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States